CLINICAL TRIAL: NCT01977781
Title: Safety and Efficacy of Topical Tacrolimus 0.05% in the Treatment of Ocular Graft-Versus-Host Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Reza Dana, MD, Principal Investigator, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-067H
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Ocular GVHD
Keywords: GVHD; Ocular GVHD; Tacrolimus; Methylprednisolone
MeSH Terms: interventions — Tacrolimus; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacrolimus (Experimental): Topical tacrolimus suspension will be formulated and aseptically prepared from commercially available intravenous tacrolimus, PROGRAF® (Astellas Pharma US, Inc), and transferred into a sterile dropper container by the MEEI pharmacy. A formulation of 0.05% (5mg/10ml) concentration of tacrolimus with diluting solvent, LiquiTears Ophthalmic Solution (Major Pharmaceuticals, Inc.) will be used. Patients will be instructed to keep refrigerated each bottle after opening for 9 days and keep frozen the unopened bottles up to 45 days. They will also be instructed to shake the bottles at least 20 times before using it.
  Interventions: Drug: Tacrolimus
- Methylprednisolone Sodium Succinate (Active Comparator): Topical methylprednisolone sodium succinate suspension will be formulated and aseptically prepared from commercially available sterile dry powder vial preservative-free for intravenous use, SOLU-MEDROL® (Pfizer, Inc.). A formulation of 0.5% (5mg/1ml) concentration of methylprednisolone with diluting solvents, LiquiTears Ophthalmic Solution (Major Pharmaceuticals, Inc.) will be used. Patients will be instructed to keep refrigerated each bottle after opening for 9 days and keep frozen the unopened bottles up to 45 days. They will also be instructed to shake the bottles at least 20 times before using it.
  Interventions: Drug: Methylprednisolone Sodium Succinate

INTERVENTIONS:
Drug: Tacrolimus — Topical bilateral application of 0.05% Tacrolimus BID for 10 weeks
  Other Names: Compounded tacrolimus (FK-506, Prograf, Protopic) in vehicle
  Arms: Tacrolimus
Drug: Methylprednisolone Sodium Succinate — Topical bilateral application of 0.5% methylprednisolone sodium succinate BID for 10 weeks
  Other Names: Compounded methlyprednisolone sodium succinate in vehicle
  Arms: Methylprednisolone Sodium Succinate

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of topical tacrolimus 0.05% twice a day in the treatment of ocular graft versus host disease (GVHD).

DETAILED DESCRIPTION:
The objective of this study is to compare the safety and efficacy of topical tacrolimus 0.05% drops compared with topical methylprednisolone sodium succinate 0.5% drops in patients with ocular GVHD. 40 patients with ocular GVHD who meet the inclusion criteria of the study as determined by a screening visit will be divided into two equal groups. In addition to their current medication, one group will receive the topical tacrolimus 0.05% drops and the other group will receive the topical methylprednisolone sodium succinate 0.5% drops. The participants will then have two follow-up visits at the week 5 and week 10 markers after their screening visit.

To evaluate the purpose of the study as well as the patient's safety, the following procedures will be performed at each visit: a comprehensive eye examination, tear break-up time (TBUT), Schirmer's test, intraocular pressure (IOP), fundoscopy and grading scores of lid margin and corneal fluorescein staining. The following questionnaires will be administered at each visit: Ocular Surface Disease Index (OSDI) and Symptom Assessment in Dry Eye (SANDE). Impression cytology specimens will be taken only at the screening visit and at the week 10 visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Willing and able to provide written informed consent.
* Willing and able to comply with study assessments for the full duration of the study.
* Diagnosis of ocular GVHD.
* Minimum corneal fluorescein staining of 4 (NEI grading scheme, 0-15) in at least one eye.
* Ocular Surface Disease Index score >22.
* In good stable overall health.

Exclusion Criteria:

* History of immune disease other than GVHD.
* Ocular or periocular malignancy.
* Significant change, as judged by the principal investigator, in systemic immunosuppressive regimen within 2 weeks of study entry.
* Any history of topical tacrolimus use.
* Any change in dosage of tetracycline compounds (tetracycline, doxycycline, and minocycline) within the last month.
* Any change in frequency of preserved anti-glaucoma medications within 2 weeks of study entry.
* Current use of topical steroids more than twice a day.
* Change in frequency of serum tears, topical cyclosporine and/or topical kineret within the last month.
* Corneal epithelial defect >1mm2.
* Any history of herpetic keratitis.
* Participation in another simultaneous medical research study.
* Signs of current infection, including fever and current treatment with antibiotics.
* Intra-ocular surgery or ocular laser surgery within 3 months.
* Pregnancy (positive pregnancy test) or lactating
* Has worn contact lenses, except for bandage contact lens or rigid gas permeable lens, for the last 2 weeks prior to the study or would be unable to stay off contact lenses for the study duration.
* Any condition (including language barrier) that precludes patient's ability to comply with study requirements including completion of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Dana, MD, MPH, MSc, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Tacrolimus: Topical tacrolimus suspension will be formulated and aseptically prepared from commercially available intravenous tacrolimus, PROGRAF® (Astellas Pharma US, Inc), and transferred into a sterile dropper container by the MEEI pharmacy. A formulation of 0.05% (5mg/10ml) concentration of tacrolimus with diluting solvent, LiquiTears Ophthalmic Solution (Major Pharmaceuticals, Inc.) will be used. Patients will be instructed to keep refrigerated each bottle after opening for 9 days and keep frozen the unopened bottles up to 45 days. They will also be instructed to shake the bottles at least 20 times before using it.
  Tacrolimus
- Methylprednisolone Sodium Succinate: Topical methylprednisolone sodium succinate suspension will be formulated and aseptically prepared from commercially available sterile dry powder vial preservative-free for intravenous use, SOLU-MEDROL® (Pfizer, Inc.). A formulation of 0.5% (5mg/1ml) concentration of methylprednisolone with diluting solvents, LiquiTears Ophthalmic Solution (Major Pharmaceuticals, Inc.) will be used. Patients will be instructed to keep refrigerated each bottle after opening for 9 days and keep frozen the unopened bottles up to 45 days. They will also be instructed to shake the bottles at least 20 times before using it.
  Methylprednisolone Sodium Succinate
Period: Overall Study
Arm/Group | Tacrolimus | Methylprednisolone Sodium Succinate
Started | 24 | 16
Completed | 18 | 15
Not Completed | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacrolimus | Methylprednisolone Sodium Succinate | Total
Number analyzed (Participants) | 24 | 16 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (11.54) | 58 (10.98) | 56 (11.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 16 | 9 | 25
Region of Enrollment [Number; unit: participants]
  United States | 24 | 16 | 40

OUTCOME MEASURES:

1. Primary Outcome: Ocular Burning Sensation, Ocular Discharge, Ocular Redness, Ocular Itching, Foreign Body Sensation
Description: Ocular burning sensation, ocular discharge, ocular redness, ocular Itching, and foreign body sensation were measured to evaluate the safety and tolerability of topical tacrolimus 0.05% twice a day in the treatment of patients with ocular GVHD. Safety and tolerability of topical tacrolimus 0.05% twice a day will be monitored by the occurrence of systemic and ocular adverse events in addition to symptoms directly related to the instillation or use of the investigational medication. Subjects will be monitored at each study visit for the occurrence of any adverse events found through examination or patient reports. Tolerability will be evaluated at every visit with a self-response questionnaire that assessed burning sensation, discharge, redness, itchiness, and foreign body sensation on a scale from 0 to 4 (none = 0, trace = 1, mild = 2, moderate = 3, and severe = 4). Where a higher value represents more symptoms (less tolerability).
Time Frame: 10 weeks
Population: The results are taken from the week 10 study assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tacrolimus | Methylprednisolone Sodium Succinate
Number analyzed (Participants) | 24 | 16
units on a scale
  Ocular Burning Sensation | 3.50 (0.98) | 2.23 (1.19)
  Ocular Discharge | 0.16 (0.51) | 0.26 (0.59)
  Ocular Redness | 1.25 (1.57) | 0.43 (0.97)
  Ocular Itching | 0.50 (0.85) | 0.60 (1.12)
  Foreign Body Sensation | 0.70 (1.29) | 0.57 (1.14)
Statistical Analysis 1: Comparison: Tacrolimus vs Methylprednisolone Sodium Succinate; Only the statistical analysis results for burning sensation at 10 weeks are reported below as they where the only tolerability results found to be significantly different between the two arms. All other tolerability measures were found to be the same between the two groups; Test type: Superiority or Other; p = 0.0019, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Ocular Surface Disease Index (OSDI) Questionnaire
Description: The OSDI questionnaire is a 12-question survey used to measure the symptoms of dry eye disease. Each of the 12 individual questions rate each of the dry eye symptoms on a 0-4 scale, with 4 meaning that the symptom is present all of the time and 0 meaning the symptom is present none of the time. The overall ODSI score is calculated by adding all of the values from the 12 questions, multiplying that value by 25, and dividing the resulting value by the number of questions answered. This results in an overall scale that ranges from 0-100, with 100 being severe dry eye symptoms and 0 being no dry eye symptoms.
Time Frame: 10 weeks
Population: Measurements are reported from the 10 week study visit. At this time 3 subjects were lost to follow-up and 4 subjects dropped out of the study due to burning sensations. 3 subjects dropped out from the Tacrolimus arm and 1 subject dropped out of the Methylprednisolone arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tacrolimus | Methylprednisolone Sodium Succinate
Number analyzed (Participants) | 18 | 15
units on a scale | 42 (20) | 28 (18)

3. Secondary Outcome: Corneal Epitheliopathy (Corneal Fluorescein Staining Using the NEI Grading Scheme)
Description: Corneal fluorescein staining is used to assess the level of corneal epitheliopathy that is related to dry eye disease. The corneal fluorescein staining scale ranges from 0 to 15, with 0 representing the minimum level of corneal epitheliopathy and 15 representing the maximum level of epitheliopathy.
Time Frame: 10 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tacrolimus | Methylprednisolone Sodium Succinate
Number analyzed (Participants) | 18 | 15
units on a scale | 3.7 (2.0) | 6.6 (3.8)

4. Secondary Outcome: Schirmer Tear Test (mm)
Description: Schirmer tear test measures the amount of tear secretion produced by a patient in millimeters (mm). Generally, the greater amounts of tear secretion is better than smaller amounts of tear secretion. The minimum value of this scale is 0 mm of tear secretion and there is no maximum value to this scale.
Time Frame: 10 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Tacrolimus | Methylprednisolone Sodium Succinate
Number analyzed (Participants) | 18 | 15
millimeter (mm) | 3.5 (2.3) | 3.5 (2.8)

5. Secondary Outcome: Tear Film Break-Up Time
Description: Tear Film Break-Up Time measures the amount of time, in seconds, that the tear film completely coats the ocular surface after each blink. The longer the amount of time the tear film completely coats the ocular surface is considered to be better than a shorter amount of time.
Time Frame: 10 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Tacrolimus | Methylprednisolone Sodium Succinate
Number analyzed (Participants) | 18 | 15
Seconds | 2.6 (3.0) | 1.0 (2.0)

6. Secondary Outcome: Visual Acuity
Description: Visual acuity is measured by asking subjects to read letters on a chart that consists of different rows of letters. Each row of letters corresponds to different levels of visual acuity. The Logarithm of the Minimum Angle of Resolution (LogMAR) scale generally ranges from 0 to 1, with 0 corresponding to 20/20 vision and 1 corresponding to 20/200 vision. The range from 0-1 is not absolute, however, as patients who have vision better than 20/20 or vision worse than 20/200 will score out side of the 0 to 1 range.
Time Frame: 10 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: LogMAR Scale
Arm/Group | Tacrolimus | Methylprednisolone Sodium Succinate
Number analyzed (Participants) | 18 | 15
LogMAR Scale | 0.13 (0.25) | 0.13 (0.20)

7. Secondary Outcome: Intraocular Pressure
Description: Intraocular pressure is the measure of the fluid pressure within the eye as measured by tonometry. Intraocular pressure is normally measured in millimeters of mercury (mmHg). The normal range for intraocular pressure is 12-20 mmHg, there is no better or worse measurement.
Time Frame: 10 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Tacrolimus | Methylprednisolone Sodium Succinate
Number analyzed (Participants) | 18 | 15
millimeters of mercury (mmHg) | 16.5 (3.6) | 17.1 (3.8)

ADVERSE EVENTS:
Time Frame: Adverse even data was collected over the entire study period, which lasted 10 weeks.
Arm/Group | Tacrolimus | Methylprednisolone Sodium Succinate
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/16
Other Adverse Events (participants affected / at risk) | 20/24 | 15/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus (N=24) | Methylprednisolone Sodium Succinate (N=16)
Ocular Burning Sensation (Eye disorders) | 18 | 15
Ocular Discharge (Eye disorders) | 18 | 15
Ocular Redness (Eye disorders) | 18 | 15
Ocular Itching (Eye disorders) | 18 | 15
Foreign Body Sensation (Eye disorders) | 17 | 14

LIMITATIONS AND CAVEATS:
This study was limited by the lack of a placebo arm, which in many dry-eye trials is characterized by a topical lubricant; however, we believe that given the disease severity among patients in this trial, inclusion of a placebo was not ethical.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No